CLINICAL TRIAL: NCT01553201
Title: The Effectiveness of Botulinum Toxin on Persistent Pelvic Pain in Women With Endometriosis
Brief Title: Botulinum Toxin for Pelvic Pain in Women With Endometriosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120083; 12-N-0083
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2018-09

CONDITIONS: Endometriosis; Chronic Pelvic Pain; Pelvic Muscle Spasm; Quality of Life
Keywords: Quality of Life; Endometriosis; Botulinum Toxin A; Pelvic Floor Muscle Spasm; Chronic Pelvic Pain
MeSH Terms: conditions — Endometriosis | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin (BoNT) (Experimental): OnabotulinumtoxinA 100 Units diluted in 4cc saline, one time intramuscular administration
  Interventions: Drug: Botulinum toxin (BoNT)
- Placebo (Placebo Comparator): Saline, 4cc, one time intramuscular administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin (BoNT) — OnabotulinumtoxinA 100 Units diluted in 4cc saline, one time intramuscular administration
  Arms: Botulinum toxin (BoNT)
Drug: Placebo — Saline, 4cc, one time intramuscular administration
  Arms: Placebo

SUMMARY:
Background:

- Some women with endometriosis have chronic pelvic pain. This pain may be caused by spasms of the pelvic floor muscles. These spasms can be detected by an examination. Studies suggest that botulinum toxin can help treat problems caused by muscle spasms. Researchers want to see if botulinum toxin injections into the pelvic floor muscles can decrease pain and spasms in women with pelvic pain.

Objectives:

- To see if botulinum toxin can relieve pain from pelvic floor spasm in women with pelvic pain.

Eligibility:

- Women between 18 and 50 years of age with pain associated with pelvic muscle spasm and endometriosis. Pain must be persistent (lasting for at least 3 months).

Design:

* Participants will keep a pain diary and record their pain medication use for a month before the first visit.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Participants will also answer questions about their pain levels and quality of life.
* Participants will receive either botulinum toxin or a placebo (salt water) injection. The injection will be given into the pelvic floor muscles through the vaginal wall. Participants will take a muscle relaxant like Valium and have anesthetic cream put on the vaginal wall before the injection.
* After the injection, participants will keep a pain diary for another month.
* At a 1-month followup visit, participants will answer questions about their pain. If the pain has not improved, all participants may have a botulinum toxin injection (no placebo) into the pelvic floor muscles as before.
* Participants will have followup visits for up to a year after the initial 1-month followup visit.

DETAILED DESCRIPTION:
Chronic pelvic pain associated with endometriosis is poorly understood. Some women with chronic pelvic pain have muscle spasm of their pelvic muscles. Muscle spasm may be a significant part of pain in women with endometriosis and other types of chronic pelvic pain. Botulinum toxin injection is widely used to treat conditions associated with excessive muscle activity and spasm. Studies of botulinum toxin injected into pelvic muscles of women with pelvic pain have shown a decrease pain and spasm, but too few women have been studied to conclude its effectiveness. We expect to show that botulinum toxin injection in women with pelvic pain will relieve some of their pelvic pain.

Eligible subjects will be otherwise healthy women who have chronic pelvic pain and a history of endometriosis. Subjects will be randomized to either botulinum toxin injection or placebo (salt water) injection. After one month, we will evaluate the presence of the pain and all women will be offered botulinum toxin injection. We will also evaluate the need for reinjection.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Female gender
* Age between 18 and 55
* History of endometriosis at surgery
* Persistent pelvic pain for at least 3 months
* Pelvic floor spasm
* Negative pregnancy test (in women who have not had a hysterectomy)
* Willing to use reliable method of contraception for the month after botulinum toxin injection including oral contraceptives, IUD, and barrier with spermicide.
* Willing and able to give informed consent
* Willing and able to comply with study requirements

EXCLUSION CRITERIA:

* Women with other causes of chronic pelvic pain including infectious, gastrointestinal, psychological disorders, fibromyalgia and chronic fatigue syndrome based on review of medical history within 1 year of first study visit,
* Untreated severe cervical dysplasia or other gynecologic condition clinically significant abnormalities on physical or laboratory examinations that require evaluation or treatment or that would make participation unsafe
* Hysterectomy and bilateral salpingo-oophorectomy
* Pregnancy
* Lactation
* Allergy to albumen or botulinum toxin
* Presence of antibodies to botulinum toxin or loss of response to previous injections for any indication
* A known neuromuscular junction disorder such as myasthenia gravis or Eaton-Lambert syndrome
* History of urinary or fecal incontinence
* Known pelvic prolapse

  * Eligibility will be based on a physical exam at NIH at the first study visit, as well as history and available medical records within 1 year before the study visit. Negative test results will be documented to confirm study eligibility. If the Pap and the GC and chlamydia tests were not done outside of the NIH within the previous year, or if documentation of the negative test results is not available, we will await the results of the screening tests done at the NIH before administering the study medication.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Karp, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbott JA, Jarvis SK, Lyons SD, Thomson A, Vancaille TG. Botulinum toxin type A for chronic pain and pelvic floor spasm in women: a randomized controlled trial. Obstet Gynecol. 2006 Oct;108(4):915-23. doi: 10.1097/01.AOG.0000237100.29870.cc. PMID 17012454
- [Background] Bhidayasiri R, Truong DD. Expanding use of botulinum toxin. J Neurol Sci. 2005 Aug 15;235(1-2):1-9. doi: 10.1016/j.jns.2005.04.017. PMID 15990116
- [Background] Jankovic J. Botulinum toxin in clinical practice. J Neurol Neurosurg Psychiatry. 2004 Jul;75(7):951-7. doi: 10.1136/jnnp.2003.034702. PMID 15201348
- [Derived] Karp BI, Tandon HK, Sinaii N, Aredo JV, Phan VT, Salmeri N, Shah JP, Merideth MA, Stratton P. Botulinum toxin for endometriosis-associated chronic pelvic pain: a randomised, double-masked, parallel, phase 2 trial. EClinicalMedicine. 2026 Jan 5;91:103740. doi: 10.1016/j.eclinm.2025.103740. eCollection 2026 Jan. PMID 41551998
- [Derived] Phan VT, Stratton P, Tandon HK, Sinaii N, Aredo JV, Karp BI, Merideth MA, Shah JP. Widespread myofascial dysfunction and sensitisation in women with endometriosis-associated chronic pelvic pain: A cross-sectional study. Eur J Pain. 2021 Apr;25(4):831-840. doi: 10.1002/ejp.1713. Epub 2021 Jan 8. PMID 33326662
- [Derived] Tandon HK, Stratton P, Sinaii N, Shah J, Karp BI. Botulinum toxin for chronic pelvic pain in women with endometriosis: a cohort study of a pain-focused treatment. Reg Anesth Pain Med. 2019 Jul 8:rapm-2019-100529. doi: 10.1136/rapm-2019-100529. Online ahead of print. PMID 31289238
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-N-0083.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin (BoNT) | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject in the placebo arm completed the study but her data was censored (i.e. not analyzed) on recommendation by the DSMB statistician, as she was one of a sister pair.
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin (BoNT) | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 10 | 13 | 23
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Pain
Description: Self reported improvement in pain symptoms - a binary measurement of improvement/no improvement
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin (BoNT) | Placebo
Number analyzed (Participants) | 15 | 14
Participants | 11 | 4

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Botulinum Toxin (BoNT) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin (BoNT) (N=15) | Placebo (N=15)
Muscular weakness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Nervous system disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT01553201/Prot_SAP_001.pdf